CLINICAL TRIAL: NCT00332397
Title: Randomized Comparison of 3 Limus Agent-Eluting Stents for the Reduction of Coronary Restenosis
Brief Title: The Efficacy of Three Different Limus Agent-Eluting Stents to Prevent Restenosis
Acronym: ISAR-TEST-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S02206
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Rapamycin-eluting Stent (Cypher)
  Interventions: Device: Rapamycin-eluting Stent
- B (Active Comparator): Zotarolimus-eluting Stent (Endeavor)
  Interventions: Device: Zotarolimus-eluting Stent
- C (Active Comparator): Rapamycin-eluting Stent
  Interventions: Device: Rapamycin-eluting Stent

INTERVENTIONS:
Device: Rapamycin-eluting Stent — due to randomization, Cypher stent will be implanted
  Other Names: Cypher
  Arms: A
Device: Zotarolimus-eluting Stent — due to randomization, Endeavor stent will be implanted
  Other Names: Endeavor
  Arms: B
Device: Rapamycin-eluting Stent — due to randomization, rapamycin-eluting stent will be implanted
  Arms: C

SUMMARY:
The purpose of this study is to evaluate the efficacy of 3 different drug-eluting-stent platforms to reduce coronary artery reblockage after stent implantation

DETAILED DESCRIPTION:
Coronary artery reblockage remains still a drawback of percutaneous coronary interventions even in the era of drug-eluting stents (DES). DESs working principle consists of the delivery of controlled amounts of antiproliferative agents at the local level, which results in the suppression of neontimal proliferation, the main cause of lumen re-narrowing after stent implantation.At present, several DES platforms have been developed and evaluated for clinical use. They differ between them with regard to the stent type, anti-proliferative drug, presence of polymers employed for drug storage and modification of drug-release kinetics as well as type of polymer used for this purpose. Most of the DES platforms have used agents from the "limus family". Although the majority of DESs employ polymer coating to control drug storage and release, in view of the increasing safety and efficacy associated with the long-term presence of polymers a strong interest has recently been shown in the development DES platforms that do not require permanent polymers. Trials as ACTION or JUPITER II have demonstrated that not all DESs are associated with the expected improved outcomes. On the other hand, not all successful DESs have been equally effective in the reduction of restenosis. Thus, rapamycin-eluting stents (Cypher stents) have been associated with lower angiographic and clinical restenosis rates than paclitaxel-eluting stents (Taxus stents). Similarly, Cypher stents have been superior to Endeavor stents regarding the primary end point of late luminal loss in the recent ENDEAVOR III trial. Meanwhile, the on-site rapamycin-coated stents (ISAR stents) had an equivalent antiproliferative efficacy to Taxus stents in the ISAR-TEST trial. However, none of these studies evaluated angiographic restenosis as their primary endpoint and no direct comparisons between the 3 DES -Cypher, Endeavor and ISAR stents, have been performed. The Cypher stent is a stainless steel stent coated with sirolimus with use of permanent polymers while the Endeavor stent is a cobalt alloy based stent coated with zotarolimus which also uses permanent polymers for drug-storage and release. The ISAR stent is a rough surface stainless steel stent that can be coated with sirolimus in the cath lab without requiring permanent polymeric coating.

ELIGIBILITY:
Inclusion Criteria:

Patients older than age 18 ´ presence of ischemic symptoms or evidence of myocardial ischemia in the presence of ≥50% de novo stenosis located in native coronary vessels written, informed consent by the patient or her/his legally-authorized representative for participation in the study.

Exclusion Criteria:

Target lesion located in the left main trunk or bypass graft In-stent restenosis Cardiogenic shock Malignancies or other comorbid conditions with life expectancy less than one year or that may result in protocol non-compliance Known allergy to the study medications: aspirin, clopidogrel, zotarolimus, sirolimus, stainless steel, or cobalt alloy Pregnancy (present, suspected or planned) or positive pregnancy test Previous enrollment in this trial Patient's inability to fully cooperate with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1007 (Actual)
Dates: Start 2006-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary end point of the study is the incidence of binary angiographic restenosis at 6-8 month follow-up angiography, measured by QCA in the in-segment area. | 6-8 months

SECONDARY OUTCOMES:
The need of target lesion revascularization defined as any revascularization procedure involving the target lesion due to luminal re-narrowing in the presence of symptoms or objective signs of ischemia. | 9-12 months
The combined incidence of death or myocardial infarction. | 9-12 months
In-stent late luminal loss. | 9-12 months
Incidence of stent thrombosis. | 9-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schoemig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - First Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Background] Mehilli J, Kastrati A, Wessely R, Dibra A, Hausleiter J, Jaschke B, Dirschinger J, Schomig A; Intracoronary Stenting and Angiographic Restenosis--Test Equivalence Between 2 Drug-Eluting Stents (ISAR-TEST) Trial Investigators. Randomized trial of a nonpolymer-based rapamycin-eluting stent versus a polymer-based paclitaxel-eluting stent for the reduction of late lumen loss. Circulation. 2006 Jan 17;113(2):273-9. doi: 10.1161/CIRCULATIONAHA.105.575977. Epub 2006 Jan 3. PMID 16391155
- [Background] Dibra A, Kastrati A, Mehilli J, Pache J, Schuhlen H, von Beckerath N, Ulm K, Wessely R, Dirschinger J, Schomig A; ISAR-DIABETES Study Investigators. Paclitaxel-eluting or sirolimus-eluting stents to prevent restenosis in diabetic patients. N Engl J Med. 2005 Aug 18;353(7):663-70. doi: 10.1056/NEJMoa044372. Epub 2005 Aug 16. PMID 16105990
- [Background] Hausleiter J, Kastrati A, Wessely R, Dibra A, Mehilli J, Schratzenstaller T, Graf I, Renke-Gluszko M, Behnisch B, Dirschinger J, Wintermantel E, Schomig A; investigators of the individualizable durg-eluting Stent System to Abrogate Restenosis Project. Prevention of restenosis by a novel drug-eluting stent system with a dose-adjustable, polymer-free, on-site stent coating. Eur Heart J. 2005 Aug;26(15):1475-81. doi: 10.1093/eurheartj/ehi405. Epub 2005 Jun 23. PMID 15975990
- [Background] Windecker S, Remondino A, Eberli FR, Juni P, Raber L, Wenaweser P, Togni M, Billinger M, Tuller D, Seiler C, Roffi M, Corti R, Sutsch G, Maier W, Luscher T, Hess OM, Egger M, Meier B. Sirolimus-eluting and paclitaxel-eluting stents for coronary revascularization. N Engl J Med. 2005 Aug 18;353(7):653-62. doi: 10.1056/NEJMoa051175. Epub 2005 Aug 16. PMID 16105989
- [Background] Serruys PW, Ormiston JA, Sianos G, Sousa JE, Grube E, den Heijer P, de Feyter P, Buszman P, Schomig A, Marco J, Polonski L, Thuesen L, Zeiher AM, Bett JH, Suttorp MJ, Glogar HD, Pitney M, Wilkins GT, Whitbourn R, Veldhof S, Miquel K, Johnson R, Coleman L, Virmani R; ACTION investigators. Actinomycin-eluting stent for coronary revascularization: a randomized feasibility and safety study: the ACTION trial. J Am Coll Cardiol. 2004 Oct 6;44(7):1363-7. doi: 10.1016/j.jacc.2004.03.084. PMID 15464314
- [Background] Kastrati A, Dibra A, Eberle S, Mehilli J, Suarez de Lezo J, Goy JJ, Ulm K, Schomig A. Sirolimus-eluting stents vs paclitaxel-eluting stents in patients with coronary artery disease: meta-analysis of randomized trials. JAMA. 2005 Aug 17;294(7):819-25. doi: 10.1001/jama.294.7.819. PMID 16106007
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Derived] Byrne RA, Kastrati A, Tiroch K, Schulz S, Pache J, Pinieck S, Massberg S, Seyfarth M, Laugwitz KL, Birkmeier KA, Schomig A, Mehilli J; ISAR-TEST-2 Investigators. 2-year clinical and angiographic outcomes from a randomized trial of polymer-free dual drug-eluting stents versus polymer-based Cypher and Endeavor [corrected] drug-eluting stents. J Am Coll Cardiol. 2010 Jun 8;55(23):2536-43. doi: 10.1016/j.jacc.2010.03.020. Epub 2010 Apr 22. PMID 20417052
- [Derived] Byrne RA, Mehilli J, Iijima R, Schulz S, Pache J, Seyfarth M, Schomig A, Kastrati A. A polymer-free dual drug-eluting stent in patients with coronary artery disease: a randomized trial vs. polymer-based drug-eluting stents. Eur Heart J. 2009 Apr;30(8):923-31. doi: 10.1093/eurheartj/ehp044. Epub 2009 Feb 24. PMID 19240066